CLINICAL TRIAL: NCT04535453
Title: A Randomized, Double-blind, Placebo-controlled Phase 2a Study to Evaluate a Range of Dose Levels and Vaccination Intervals of Ad26.COV2.S in Healthy Adults Aged 18 to 55 Years Inclusive and Adults Aged 65 Years and Older and to Evaluate 2 Dose Levels of Ad26.COV2.S in Healthy Adolescents Aged 12 to 17 Years Inclusive
Brief Title: A Study to Evaluate a Range of Dose Levels and Vaccination Intervals of Ad26.COV2.S in Healthy Adults and Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR108854; VAC31518COV2001 (Other: Janssen Vaccines & Prevention B.V.); 2020-002584-63 (EudraCT Number)
Expanded Access: NCT04817657 (No longer available)
Record Dates: First submitted 2020-08-27; First posted 2020-09-02 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Healthy
MeSH Terms: interventions — Ad26COVS1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Groups 1-6 (Experimental): Participants will receive a 2-dose Ad26.COV2.S vaccination regimen at Days 1 and 57 at different dose levels (Groups 1-3), or a single-dose Ad26.COV2.S vaccination regimen at different dose levels (Groups 4-5), or placebo (Group 6). At unblinded phase, participants in Group 6 initially receiving placebo will be offered 2 doses of Ad26.COV2.S vaccine at a single dose level, at a 28-day interval. Participants will also receive a single antigen presentation injection with single dose level of Ad26.COV2.S at 4 months after second vaccination (Groups 1-5) or placebo (Group 6).
  Interventions: Biological: Ad26.COV2.S; Other: Placebo
- Groups 7-8 (Experimental): Participants will receive 2-dose Ad26.COV2.S vaccination regimen at Days 1 and 29 at fixed dose level (Groups 7) or placebo (Groups 8). At unblinded phase, participants in Group 8 initially receiving placebo will be offered 2 doses of Ad26.COV2.S vaccine at a single dose level, at a 28-day interval. Participants will also receive a single antigen presentation injection with single dose level of Ad26.COV2.S at 4 months after second vaccination (Group 7) or placebo (Group 8).
  Interventions: Biological: Ad26.COV2.S; Other: Placebo
- Groups 9-10 (Experimental): Participants will receive 2-dose Ad26.COV2.S vaccination regimen at Days 1 and 85 at fixed dose level (Group 9) or placebo (Group 10). At unblinded phase, participants in Group 10 initially receiving placebo will be offered 2 doses of Ad26.COV2.S vaccine at a single dose level, at a 28-day interval. Participants will also receive a single antigen presentation injection with single dose level of Ad26.COV2.S at 4 months after second vaccination (Group 9) or placebo (Group 10).
  Interventions: Biological: Ad26.COV2.S; Other: Placebo
- Groups A-C (Experimental): Participants will receive a single dose Ad26.COV2.S vaccination regimen at Day 1 at fixed dose level (Groups A and B) or placebo (Group C). At approximately 6 months of study participation (unblinded phase), participants in Group C initially receiving placebo will receive Ad26.COV2.S vaccine at a single dose level, at a 56-day interval.
  Interventions: Biological: Ad26.COV2.S; Other: Placebo

INTERVENTIONS:
Biological: Ad26.COV2.S — All participants, both adults and adolescents, will receive intramuscular (IM) injections of Ad26.COV2.S.
  Other Names: JNJ-78436735, Ad26COVS1
Other: Placebo — Adult participants in Groups 4, 5, 6, 8, and 10, and adolescent participants in Group C will receive at least one injection of placebo.

SUMMARY:
The primary purpose of this study is to assess humoral immune responses of 3 dose levels of Ad26.COV2.S administered intramuscularly (IM) as a 2-dose schedule (56 days apart); Ad26.COV2.S administered IM as a single vaccination; safety and reactogenicity of Ad26.COV2.S administered IM as a 2-dose or a single-dose schedule in adults (18-65 years or older) and to assess the safety and reactogenicity of Ad26.COV2.S, administered IM as single dose in adolescents (12-17 years) and to test both compressed and expanded 2-dose schedules of Ad26.COV2.S (28 and 84 days apart) in adults (18-55 years and 65 years or older).

DETAILED DESCRIPTION:
The aim of the COVID-19 vaccine clinical development program is to develop a safe and effective vaccine for the prevention of COVID-19. Currently, there is only limited availability of authorized/licensed vaccines for the prevention of coronavirus disease-2019 (COVID-19). Ad26.COV2.S (also known as Ad26COVS1) is a monovalent vaccine composed of a recombinant, replication incompetent adenovirus type 26 (Ad26) vector, constructed to encode the severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) virus spike (S) protein, which will be assessed in this study. Also, different vaccination intervals and multiple lower dose levels compared to the dose levels in the first in human study (VAC31518COV1001 [NCT04436276]) will be assessed. For adults, the study consists of: screening phase (28 days), vaccination phase (1-3 months) depending on the vaccination interval, and follow-up (12 months). The study duration is approximately 15 months (Groups 1-6, 8, 10 and Group 7 [to participants for whom vaccination 2 was delayed]), 14 months (Group 7), and 16 months (Group 9) in adult groups and approximately 13 months for adolescents group (Groups A to C). The adverse events and other safety assessments including vital signs measurements (heart rate, supine systolic and diastolic blood pressure, respiratory rate, and body temperature), and physical examinations will be assessed during the study.

Note: The Informed Consent Form dated 27-Oct-2020 is final version of the study MASTER ICF, used by local countries to prepare the local language version of the ICF, which have been approved by the Ethics Committees.

And the highlighted text in the ICF document are the guidance for country specific adaptation.

ELIGIBILITY:
Inclusion Criteria:

For Adults

* Participant must have a body mass index (BMI) less than (<) 30.0 kilogram per meter square (kg/m^2)
* Participant is 18 to 55 years of age, inclusive, or 65 years of age or older on the day of signing the informed consent form (ICF).
* Participant 18 to 55 years of age, inclusive: participant must be healthy, in the investigator's clinical judgment, as confirmed by medical history, physical examination, and vital signs performed at screening, and must not have comorbidities related to an increased risk of severe coronavirus disease-2019 (COVID-19), except for smoking and mild hypertension, which are allowed. Participant 65 years of age and older: In the investigator's clinical judgment, participant must be either in good or stable health. Participant may have underlying illnesses, as long as the symptoms and signs are medically controlled and not considered to be comorbidities related to an increased risk of severe COVID-19, except for smoking and mild hypertension, which are allowed. If on medication for a condition, the medication dose must have been stable for at least 12 weeks preceding vaccination and expected to remain stable for the duration of the study. Participant will be included on the basis of physical examination, medical history, and vital signs
* Participant will be included on the basis of physical examination, medical history, and vital signs
* All participants of childbearing potential must: a) Have a negative highly sensitive urine pregnancy test at screening, b)Have a negative highly sensitive urine pregnancy test immediately prior to each study vaccine administration
* Participant agrees to not donate bone marrow, blood, and blood products from the first study vaccine administration until 3 months after receiving the last dose of study vaccine
* Participant must be willing to provide verifiable identification, has means to be contacted and to contact the investigator during the study

For Adolescents:

* Participant is 12 to 17 years of age, inclusive, on the day of signing the informed consent form (ICF)
* Participants must have signed an ICF (or their legally acceptable representative or parent(s) [preferably both parents if available or as per local requirements] must sign) indicating that they understand the purpose of, and procedures required for, the study, are willing/able to adhere to the prohibitions and restrictions specified in the protocol and study procedures, and are willing (or the parents are willing for their adolescent) to participate in the study. Informed assent must be obtained from adolescents, depending on local regulations and practice
* Participant must be healthy, in the investigator's clinical judgment, as confirmed by medical history, physical examination, and vital signs performed at screening, and must not have comorbidities related to an increased risk of severe COVID-19

Exclusion Criteria:

For Adults

* Participant has a clinically significant acute illness (this does not include minor illnesses such as diarrhea or mild upper respiratory tract infection) or temperature greater than or equal to (>=) 38.0 degree Celsius [C] (100.4 degree Fahrenheit [F]) within 24 hours prior to the planned first dose of study vaccine; randomization at a later date is permitted at the discretion of the investigator and after consultation with the sponsor
* Participant has a history of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which is considered cured with minimal risk of recurrence)
* Participant has a known or suspected allergy or history of anaphylaxis or other serious adverse reactions to vaccines or their excipients (including specifically the excipients of the study vaccine)
* Participant received treatment with immunoglobulins in the 3 months or blood products in the 4 months before the planned administration of the first dose of study vaccine or has any plans to receive such treatment during the study
* Participant received an investigational drug (including investigational drugs for prophylaxis of COVID-19) or used an invasive investigational medical device within 30 days or received investigational Ig or monoclonal antibodies within 3 months, or received convalescent serum for COVID-19 treatment within 4 months or received an investigational vaccine (including investigational Adenoviral-vectored vaccines) within 6 months before the planned administration of the first dose of study vaccine or is currently enrolled or plans to participate in another investigational study during the course of this study For Adolescents
* Participant has a known or suspected allergy or history of anaphylaxis or other serious adverse reactions to vaccines or their excipients (including specifically the excipients of the study vaccine)
* Participants with a history of illness or with an ongoing illness that, in the opinion of the investigator, may pose additional risk to the participant if he/she participates in the study
* Participant has a history of Kawasaki disease
* Participant has a history of an underlying clinically significant acute or chronic medical condition or physical examination findings for which, in the opinion of the investigator, participation would not be in the best interest of the participant (example, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 635 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (13):
- Germany (3):
  - Charité Research Organisation GmbH, Berlin
  - CTC North GmbH & Co. KG, Am Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitaetsmedizin Rostock, Rostock
- Netherlands (3):
  - PRA Health Sciences, Groningen
  - Centre for Human Drug Research, Leiden
  - UMCU, Utrecht
- Spain (3):
  - Hosp. Univ. de La Princesa, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp. Univ. Marques de Valdecilla, Santander
- United Kingdom (4):
  - Alder Hey Hospital, Liverpool
  - St George's, University of London, London
  - Royal Manchester Children's Hospital, Manchester
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Cardenas V, Le Gars M, Truyers C, Ruiz-Guinazu J, Struyf F, Colfer A, Bonten M, Borobia A, Reisinger EC, Kamerling IMC, Douoguih M, Sadoff J. Safety and immunogenicity of Ad26.COV2.S in adults: A randomised, double-blind, placebo-controlled Phase 2a dose-finding study. Vaccine. 2024 Jun 11;42(16):3536-3546. doi: 10.1016/j.vaccine.2024.04.059. Epub 2024 May 4. PMID 38705804
- [Derived] Sadoff J, Le Gars M, Brandenburg B, Cardenas V, Shukarev G, Vaissiere N, Heerwegh D, Truyers C, de Groot AM, Jongeneelen M, Kaszas K, Tolboom J, Scheper G, Hendriks J, Ruiz-Guinazu J, Struyf F, Van Hoof J, Douoguih M, Schuitemaker H. Durable antibody responses elicited by 1 dose of Ad26.COV2.S and substantial increase after boosting: 2 randomized clinical trials. Vaccine. 2022 Jul 30;40(32):4403-4411. doi: 10.1016/j.vaccine.2022.05.047. Epub 2022 Jun 3. PMID 35667914

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 635 participants were randomized, of which 617 were vaccinated and included in the analysis. As planned, combined data of Adolescents Groups A and B was collected and reported throughout the study.
Groups:
- Group 1: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp: Adult participants received 2-dose regimen intramuscular (IM) injection of Ad26.COV2.S vaccine at a dose level of 5*10^10 virus particles (vp) on Days 1 and 57. Participants also received a single antigen presentation IM injection of Ad26.COV2.S 1.25*10^10 vp at 4 months after second vaccination.
- Group 2: Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp: Adult participants received 2-dose regimen IM injection of Ad26.COV2.S vaccine at dose level of 2.5*10^10 vp on Days 1 and 57. Participants also received a single antigen presentation IM injection of Ad26.COV2.S 1.25*10^10 vp at 4 months after second vaccination.
- Group 3: Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp: Adult participants received 2-dose regimen IM injection of Ad26.COV2.S vaccine at dose level of 1.25*10^10 vp on Days 1 and 57. Participants also received a single antigen presentation IM injection of Ad26.COV2.S 1.25*10^10 vp at 4 months after second vaccination.
- Group 4: Ad26.COV2.S 1*10^11 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp: Adult participants received single dose regimen IM injection of Ad26.COV2.S vaccine at dose level of 1*10^11 vp on Day 1 and placebo at Day 57. Participants also received a single antigen presentation IM injection of Ad26.COV2.S 1.25*10^10 vp at 4 months after second vaccination.
- Group 5: Ad26.COV2.S 5*10^10 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp: Adult participants received a single dose regimen IM injection of Ad26.COV2.S vaccine at dose level of 5*10^10 vp on Day 1 and placebo at Day 57. Participants also received a single antigen presentation IM injection of Ad26.COV2.S 1.25*10^10 vp at 4 months after second vaccination.
- Group 6: Placebo, Placebo, Placebo: Adult participants received IM injection of placebo matching to Ad26.COV2.S vaccine on Days 1 and 57. Participants also received a single antigen presentation IM injection with single dose level of placebo matching to Ad26.COV2.S at 4 months after second vaccination. With the implementation of Amendment 5, Adults who received placebo in the primary vaccine regimen received a 2-dose active Ad26.COV2.S 5*10^10 vp IM injection vaccine regimen at a 28-day interval.
- Group 7: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp: Adult participants received 2 dose regimen IM injection of Ad26.COV2.S vaccine at dose level of 5*10^10 vp on Days 1 and 29. Participants also received a single antigen presentation IM injection of Ad26.COV2.S 1.25*10^10 vp at 4 months after second vaccination.
- Group 8: Placebo, Placebo, Placebo: Adult participants received IM injection of placebo matching to Ad26.COV2.S vaccine on Days 1 and 29. Participants also received a single antigen presentation IM injection of placebo matching to Ad26.COV2.S at 4 months after second vaccination. With the implementation of Amendment 5, adults who received placebo in the primary vaccine regimen received a 2-dose active Ad26.COV2.S vaccine regimen at a 28-day interval and at a dose level of 5*10^10 vp.
- Group 9: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp: Adult participants received 2 dose regimen IM injection of Ad26.COV2.S vaccine at dose level of 5*10^10 vp on Days 1 and 85. Participants also received a single antigen presentation injection of Ad26.COV2.S 1.25*10^10 vp at 4 months after second vaccination.
- Group 10: Placebo, Placebo, Placebo: Adult participants received IM injection of placebo matching to Ad26.COV2.S vaccine on Days 1 and 85. Participants also received a single antigen presentation IM injection of placebo matching to Ad26.COV2.S at 4 months after second vaccination. With the implementation of Amendment 5, adults who received placebo in the primary vaccine regimen received a 2-dose active Ad26.COV2.S vaccine regimen at a 28-day interval and at a dose level of 5*10^10 vp.
- Group A and B Combined: Ad26.COV2.S 2.5*10^10: Adolescent participants aged 16 to 17 years received single dose IM injection of Ad26.COV2.S vaccine at a dose level of 2.5*10^10 vp on Day 1 in Groups A and B.
- Group C: Placebo: Adolescent participants aged 16 to 17 years received single dose IM injection of placebo matching to Ad26.COV2.S vaccine on Day 1. At approximately 6 months of study participation, participants were unblinded and received vaccination 1 with Ad26.COV2.S 2.5*10^10 vp.
Period: Overall Study
Arm/Group | Group 1: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 2: Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 3: Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 4: Ad26.COV2.S 1*10^11 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 5: Ad26.COV2.S 5*10^10 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 6: Placebo, Placebo, Placebo | Group 7: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 8: Placebo, Placebo, Placebo | Group 9: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 10: Placebo, Placebo, Placebo | Group A and B Combined: Ad26.COV2.S 2.5*10^10 | Group C: Placebo
Started | 86 | 81 | 75 | 74 | 81 | 26 | 56 | 27 | 53 | 25 | 30 | 3
Completed | 82 | 73 | 70 | 70 | 75 | 24 | 54 | 25 | 50 | 23 | 30 | 2
Not Completed | 4 | 8 | 5 | 4 | 6 | 2 | 2 | 2 | 3 | 2 | 0 | 1
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0 | 3 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 6 | 3 | 3 | 2 | 1 | 1 | 1 | 1 | 1 | 0 | 1
Not completed — Other | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 2: Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 3: Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 4: Ad26.COV2.S 1*10^11 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 5: Ad26.COV2.S 5*10^10 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 6: Placebo, Placebo, Placebo | Group 7: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 8: Placebo, Placebo, Placebo | Group 9: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 10: Placebo, Placebo, Placebo | Group A and B Combined: Ad26.COV2.S 2.5*10^10 | Group C: Placebo | Total
Number analyzed (Participants) | 86 | 81 | 75 | 74 | 81 | 26 | 56 | 27 | 53 | 25 | 30 | 3 | 617
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (18.12) | 49.1 (19.44) | 49.2 (17.33) | 50.3 (17.1) | 48.6 (18.5) | 48.4 (16.88) | 48.8 (17.15) | 49.0 (17.63) | 48.1 (18.99) | 52.4 (13.63) | 16.3 (0.47) | 16.3 (0.58) | 47.4 (18.81)
Age, Customized [Count of Participants; unit: Participants]
  Children (2-11 years) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Adolescents (16-17 years) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 30 | 3 | 33
  Adults (18-64 years) | 57 | 48 | 52 | 48 | 51 | 16 | 37 | 17 | 33 | 16 | 0 | 0 | 375
  From 65 to 84 years | 29 | 33 | 23 | 26 | 30 | 10 | 19 | 10 | 20 | 9 | 0 | 0 | 209
  85 years and over | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 30 | 22 | 32 | 35 | 13 | 14 | 10 | 19 | 13 | 20 | 2 | 236
  Male | 60 | 51 | 53 | 42 | 46 | 13 | 42 | 17 | 34 | 12 | 10 | 1 | 381
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 22 | 20 | 20 | 22 | 8 | 14 | 6 | 9 | 6 | 0 | 0 | 149
  Not Hispanic or Latino | 61 | 56 | 51 | 51 | 58 | 17 | 40 | 18 | 41 | 18 | 29 | 2 | 442
  Unknown or Not Reported | 3 | 3 | 4 | 3 | 1 | 1 | 2 | 3 | 3 | 1 | 1 | 1 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Asian | 0 | 0 | 2 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 4
  White | 83 | 76 | 71 | 73 | 79 | 25 | 55 | 27 | 53 | 24 | 29 | 3 | 598
  More than one race | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Adults of Groups 1, 2 and 3: Percentage of Participants With Serological Response to Vaccination as Measured by Virus Neutralization Assay (VNA) Titers at 28 Days After Vaccination 2
Description: Percentage of participants with serological response to vaccination as measured by VNA titers were reported. A participant was considered a responder if at least one of the following conditions was met: 1) The baseline sample value was less than or equal to the lower limit of quantification (<=LLOQ) and the post-baseline sample was greater than (>) LLOQ. 2) The baseline sample value was >LLOQ and the post-baseline sample value represented an at least 4-fold (greater than or equal to [>=] 4-fold) increase from the baseline sample value. The lower limit and upper limit of quantification were 50 percent (%) inhibitory concentration (IC50) of 58 and 12,800 international unit per milliliter (IU/mL) respectively.
Time Frame: 28 days after Vaccination 2 (Day 85)
Population: Per protocol immunogenicity (PPI) set included all randomized and vaccinated participants with immunogenicity data available excluding participants with major protocol deviations expected to impact immunogenicity outcomes. Samples obtained after missed vaccinations or participants with natural SARS-CoV-2 infection (positive PCR test or N-serology) after screening were excluded from analysis. N(Overall number of participants analyzed) signifies participants evaluated for this outcome measure(OM).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 2: Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 3: Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp
Number analyzed (Participants) | 31 | 36 | 36
Percentage of participants | 96.8 (83.3) [83.3 to 99.9] | 100.0 (90.3) [90.3 to 100.0] | 88.9 (73.9) [73.9 to 96.9]

2. Primary Outcome: Adults of Groups 1, 2 and 3: Percentage of Participants With Serological Response to Vaccination as Measured by Spike Binding Antibodies Enzyme-linked Immunosorbent Assay (S-ELISA) at 28 Days After Vaccination 2
Description: Percentage of participants with serological response to vaccination as measured by S-ELISA were reported. A participant was considered a responder if at least one of the following conditions was met: 1) The baseline sample value was <=LLOQ and the post-baseline sample was >LLOQ. 2) The baseline sample value was >LLOQ and the post-baseline sample value represented an at least 4-fold (>= 4-fold) increase from the baseline sample value. The lower limit and upper limit of quantification were IC50 of 58 and 12,800 IU/mL respectively.
Time Frame: 28 days after Vaccination 2 (Day 85)
Population: PPI set included all randomized and vaccinated participants with immunogenicity data available excluding participants with major protocol deviations expected to impact immunogenicity outcomes. Samples obtained after missed vaccinations or participants with natural SARS-CoV-2 infection (defined as a positive PCR test or positive N-serology) occurring after screening were excluded from the analysis. Here, 'N' (overall number of participants analyzed) signifies participants evaluated for this OM.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 2: Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 3: Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp
Number analyzed (Participants) | 68 | 67 | 60
Percentage of participants | 100.0 (94.7) [94.7 to 100.0] | 100.0 (94.6) [94.6 to 100.0] | 96.7 (88.5) [88.5 to 99.6]

3. Primary Outcome: Adults of Groups 1, 2 and 3: Antibody Geometric Mean Titers (GMTs) as Measured by VNA at 28 Days After Vaccination 2
Description: Antibody GMTs as measured by VNA at 28 days after Vaccination 2 were reported.
Time Frame: 28 days after Vaccination 2 (Day 85)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 2: Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 3: Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp
Number analyzed (Participants) | 32 | 36 | 37
Titer | 455 (321) [321 to 645] | 490 (376) [376 to 637] | 364 (239) [239 to 556]

4. Primary Outcome: Adults of Groups 1, 2 and 3: Antibody Geometric Mean Concentrations (GMCs) as Measured by (S-ELISA) at 28 Days After Vaccination 2
Description: Antibody GMCs as measured by S-ELISA at 28 days after Vaccination 2 were reported.
Time Frame: 28 days after Vaccination 2 (Day 85)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA unit per milliliter (EU/mL)
Arm/Group | Group 1: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 2: Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 3: Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp
Number analyzed (Participants) | 71 | 68 | 60
ELISA unit per milliliter (EU/mL) | 1742 (1400) [1400 to 2168] | 1563 (1273) [1273 to 1918] | 1130 (802) [802 to 1593]

5. Primary Outcome: Adults of Groups 4, 5 and 6: Percentage of Participants With Serological Response to Vaccination as Measured by VNA Titers at 28 Days After Vaccination 1
Description: Percentage of participants with serological response to vaccination as measured by VNA titers were reported. A participant was considered a responder if at least one of the following conditions was met: 1) The baseline sample value was <=LLOQ and the post-baseline sample was >LLOQ. 2) The baseline sample value was >LLOQ and the post-baseline sample value represented an at least 4-fold (>= 4-fold) increase from the baseline sample value. The lower limit and upper limit of quantification were IC50 of 58 and 12,800 IU/mL respectively.
Time Frame: 28 days after Vaccination 1 (Day 29)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 4: Ad26.COV2.S 1*10^11 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 5: Ad26.COV2.S 5*10^10 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 6: Placebo, Placebo, Placebo
Number analyzed (Participants) | 37 | 34 | 14
Percentage of participants | 97.3 (85.8) [85.8 to 99.9] | 100.0 (89.7) [89.7 to 100.0] | 0.0 (0.0) [0.0 to 23.2]

6. Primary Outcome: Adults of Groups 4, 5 and 6: Percentage of Participants With Serological Response to Vaccination as Measured by S-ELISA at 28 Days After Vaccination 1
Description: as for outcome 2
Time Frame: 28 days after Vaccination 1 (Day 29)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 4: Ad26.COV2.S 1*10^11 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 5: Ad26.COV2.S 5*10^10 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 6: Placebo, Placebo, Placebo
Number analyzed (Participants) | 65 | 65 | 19
Percentage of participants | 98.5 (91.7) [91.7 to 100.0] | 95.4 (87.1) [87.1 to 99.0] | 0.0 (0.0) [0.0 to 17.6]

7. Primary Outcome: Adults of Groups 4, 5 and 6: Antibody GMTs as Measured by VNA at 28 Days After Vaccination 1
Description: Antibody GMTs as measured by VNA at 28 days after vaccination 1 were reported. LLOQ was 58 IU/mL.
Time Frame: 28 days after Vaccination 1 (Day 29)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 4: Ad26.COV2.S 1*10^11 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 5: Ad26.COV2.S 5*10^10 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 6: Placebo, Placebo, Placebo
Number analyzed (Participants) | 37 | 35 | 14
Titer | 263 [201 to 345] | 253 [207 to 308] | NA [NA to NA] — Geometric mean' and 95% 'confidence interval' could not be estimated as the analyzed values were below the LLOQ.

8. Primary Outcome: Adults of Groups 4, 5 and 6: Antibody GMCs as Measured by S-ELISA 28 Days After Vaccination 1
Description: Antibody GMCs as measured by S-ELISA at 28 days after Vaccination 1 were reported. The LLOQ was 50.3 IU/mL.
Time Frame: 28 days after Vaccination 1 (Day 29)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group 4: Ad26.COV2.S 1*10^11 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 5: Ad26.COV2.S 5*10^10 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 6: Placebo, Placebo, Placebo
Number analyzed (Participants) | 66 | 65 | 19
EU/mL | 505 [415 to 614] | 360 [276 to 471] | NA [NA to NA] — Geometric mean' and 95% 'confidence interval' could not be estimated as the analyzed values were below the LLOQ

9. Primary Outcome: Adults of Groups 9 and 10: Percentage of Participants With Serological Response to Vaccination as Measured by VNA Titers 28 Days After Vaccination 2
Description: as for outcome 5
Time Frame: 28 days after Vaccination 2 ( Day 113)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 9: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 10: Placebo, Placebo, Placebo
Number analyzed (Participants) | 35 | 13
Percentage of participants | 100.0 (90.0) [90.0 to 100.0] | 15.4 (1.9) [1.9 to 45.4]

10. Primary Outcome: Adults of Groups 9 and 10: Percentage of Participant With Serological Response to Vaccination as Measured by S-ELISA at 28 Days After Vaccination 2
Description: Percentage of participant with serological response to vaccination as measured by S-ELISA were reported. A participant was considered a responder if at least one of the following conditions was met: 1) The baseline sample value was <=LLOQ and the post-baseline sample was >LLOQ. 2) The baseline sample value was >LLOQ and the post-baseline sample value represented an at least 4-fold (>= 4-fold) increase from the baseline sample value. The lower limit and upper limit of quantification were IC50 of 58 and 12,800 IU/mL respectively.
Time Frame: 28 days after Vaccination 2 (Day 113)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 9: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 10: Placebo, Placebo, Placebo
Number analyzed (Participants) | 46 | 23
Percentage of participants | 100.0 (92.3) [92.3 to 100.0] | 4.3 (0.1) [0.1 to 21.9]

11. Primary Outcome: Adults of Groups 9 and 10: Antibody GMTs as Measured by VNA at 28 Days After Vaccination 2
Description: Antibody GMTs as measured by VNA at 28 days after Vaccination 2 were reported. The LLOQ was 58 IU/mL.
Time Frame: 28 days after Vaccination 2 (Day 113)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 9: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 10: Placebo, Placebo, Placebo
Number analyzed (Participants) | 35 | 13
Titer | 901 [686 to 1185] | NA [NA to NA] — Geometric mean' and 95%'confidence interval' could not be estimated as the analyzed values were below the LLOQ.

12. Primary Outcome: Adults of Groups 9 and 10: Antibody GMCs as Measured by S-ELISA at 28 Days After Vaccination 2
Description: Antibody GMCs as measured by S-ELISA at 28 days after Vaccination 2 were reported. The LLOQ was 50.3 IU/mL.
Time Frame: 28 Days after Vaccination 2 (Day 113)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group 9: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 10: Placebo, Placebo, Placebo
Number analyzed (Participants) | 46 | 23
EU/mL | 2391 [1811 to 3156] | NA [NA to NA] — 'Geometric mean' and 95% 'confidence interval' could not be estimated as the analyzed values were below the LLOQ.

13. Primary Outcome: Adults of Groups 2 to 5, Group 9-10, 1 and 7 Combined, 6 and 8 Combined: Number of Participants With Solicited Local Adverse Events (AEs) for 7 Days After Vaccination 1
Description: Number of participants with solicited local AEs at 7 days after vaccination 1 were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local AEs were pre-defined local (at the injection site) AEs for which participants were specifically questioned and which were noted by participants in their e-diary for 7 days after vaccination 1 (day of vaccination and the subsequent 7 days). Solicited local AEs included: injection site pain/tenderness, erythema and swelling at the vaccination site.
Time Frame: 7 days after Vaccination 1 (Day 8)
Population: FAS included all participants with at least one vaccine administration documented. Here, 'N' (Overall number of participants analyzed) signifies participants evaluated for this outcome measure. Participants from Groups 7 and 8 (with vaccination 2 delayed due to pausing rule) were analyzed with Groups 1 and 6, respectively in FAS for this OM. Hence, combined data for Groups 1 and 7, and Groups 6 and 8 was reported.
Measure: Count of Participants; unit: Participants
Groups:
- Groups 1 and 7 Combined: Adult participants received 2-dose regimen IM injection of Ad26.COV2.S vaccine at a dose level of 5*10^10 vp on Days 1 and 57 and also received a single antigen presentation IM injection of Ad26.COV2.S at 1.25*10^10 vp at 4 months after second vaccination.
- Group 6 and 8 Combined: Adult participants received IM injection of Ad26.COV2.S vaccine matching placebo on Days 1 and 57 and also received a single antigen presentation IM injection with single dose level of placebo matching to Ad26.COV2.S at 4 months after second vaccination.
Arm/Group | Group 2: Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 3: Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 4: Ad26.COV2.S 1*10^11 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 5: Ad26.COV2.S 5*10^10 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 9: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 10: Placebo, Placebo, Placebo | Groups 1 and 7 Combined | Group 6 and 8 Combined
Number analyzed (Participants) | 81 | 75 | 74 | 81 | 53 | 25 | 141 | 52
Participants | 27 | 24 | 39 | 42 | 21 | 2 | 75 | 7

14. Primary Outcome: Adults of Groups 2 to 5, Group 9-10, 1 and 7 Combined, 6 and 8 Combined: Number of Participants With Solicited Systemic Adverse Events (AEs) for 7 Days After Vaccination 1
Description: Number of participants with solicited systemic AEs at 7 days after vaccination 1 were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Participants were instructed on how to note signs and symptoms in their diary on a daily basis for 7 days post-vaccination (Day of vaccination and the subsequent 7 days) for solicited systemic AEs. Solicited systemic AEs included fatigue, headache, myalgia, nausea and fever (body temperature greater than or equal to [>=] 38 degree Celsius).
Time Frame: 7 days after Vaccination 1 (Day 8)
Population: FAS included all participants with at least one vaccine administration documented. Here, 'N' (Overall number of participants analyzed) signifies participants evaluated for this outcome measure. Participants from Groups 7 and 8 (with vaccination 2 delayed due to pausing rule) were analyzed with Groups 1 and 6, respectively in FAS for this OM. Hence, combined data for Groups 1 and 7, and Groups 6 and 8 is reported.
Measure: Count of Participants; unit: Participants
Groups:
- Group 1 and 7 Combined: Adult participants received 2-dose regimen IM injection of Ad26.COV2.S vaccine at a dose level of 5*10^10 vp on Days 1 and 57 and also received a single antigen presentation IM injection of Ad26.COV2.S at 1.25*10^10 vp at 4 months after second vaccination.
- Group 6 and 8 Combined: Adult subjects received IM injection of Ad26.COV2.S vaccine matching placebo on Days 1 and 57 and also received a single antigen presentation IM injection with single dose level of placebo matching to Ad26.COV2.S at 4 months after second vaccination.
Arm/Group | Group 2: Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 3: Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 4: Ad26.COV2.S 1*10^11 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 5: Ad26.COV2.S 5*10^10 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 9: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 10: Placebo, Placebo, Placebo | Group 1 and 7 Combined | Group 6 and 8 Combined
Number analyzed (Participants) | 81 | 75 | 74 | 81 | 53 | 25 | 141 | 52
Participants | 35 | 31 | 56 | 50 | 32 | 10 | 84 | 18

15. Primary Outcome: Adults of Groups 2 to 5, Group 9-10, 1 and 7 Combined, 6 and 8 Combined: Number of Participants With Solicited Local AEs at 7 Days After Vaccination 2
Description: Number of participants with solicited local AEs at 7 days after vaccination 2 were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local AEs were pre-defined local (at the injection site) AEs for which participants were specifically questioned and which were noted by participants in their e-diary for 7 days post vaccination 2 (day of vaccination and the subsequent 7 days). Solicited local AEs included: injection site pain/tenderness, erythema and swelling at the vaccination site.
Time Frame: 7 days after Vaccination 2 (Day 64 for Groups 1-6; Day 92 for Groups 9 and 10)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 3: Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 4: Ad26.COV2.S 1*10^11 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 5: Ad26.COV2.S 5*10^10 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 9: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 10: Placebo, Placebo, Placebo | Group 1 and 7 Combined | Group 6 and 8 Combined
Number analyzed (Participants) | 81 | 75 | 74 | 81 | 53 | 25 | 141 | 52
Participants | 33 | 29 | 5 | 4 | 20 | 2 | 63 | 3

16. Primary Outcome: Adults of Groups 2 to 5, Group 9-10, 1 and 7 Combined, 6 and 8 Combined: Number of Participants With Solicited Systemic AEs at 7 Days After Vaccination 2
Description: Number of participants with solicited systemic AEs at 7 days after vaccination 2 were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Participants were instructed on how to note signs and symptoms in their diary on a daily basis for 7 days post-vaccination 2 (Day of vaccination 2 and the subsequent 7 days) for solicited systemic AEs. Solicited systemic AEs included fatigue, headache, myalgia, nausea and fever (body temperature greater than or equal to [>=] 38 degree Celsius).
Time Frame: 7 days after Vaccination 2 (Day 64 for Group 1-6; Day 92 for Group 9 and 10)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 3: Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 4: Ad26.COV2.S 1*10^11 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 5: Ad26.COV2.S 5*10^10 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 9: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 10: Placebo, Placebo, Placebo | Group 1 and 7 Combined | Group 6 and 8 Combined
Number analyzed (Participants) | 81 | 75 | 74 | 81 | 53 | 25 | 141 | 52
Participants | 32 | 25 | 24 | 20 | 26 | 6 | 81 | 14

17. Primary Outcome: Adults of Groups 2 to 5, Group 9-10, 1 and 7 Combined, 6 and 8 Combined: Number of Participants With Unsolicited AEs at 28 Days After Vaccination 1
Description: Unsolicited AEs were all AEs for which the participants were not specifically questioned in the participant diary.
Time Frame: 28 days after Vaccination 1 (Day 29)
Population: FAS included all participants with at least one vaccine administration documented. Here, 'N' (Overall number of participants analyzed) signifies participants evaluated for this outcome measure. Participants from groups 7 and 8 (with vaccination 2 delayed due to pausing rule) were analyzed with groups 1 and 6 in FAS for this OM. Hence, combined data for Groups 1 and 7, and Groups 6 and 8 is reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 3: Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 4: Ad26.COV2.S 1*10^11 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 5: Ad26.COV2.S 5*10^10 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 9: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 10: Placebo, Placebo, Placebo | Group 1 and 7 Combined | Group 6 and 8 Combined
Number analyzed (Participants) | 81 | 75 | 74 | 81 | 53 | 25 | 141 | 52
Participants | 25 | 15 | 33 | 30 | 8 | 5 | 39 | 9

18. Primary Outcome: Adults of Groups 2 to 5, Group 9-10, 1 and 7 Combined, 6 and 8 Combined: Number of Participants With Unsolicited AEs at 28 Days After Vaccination 2
Description: Unsolicited AEs were all AEs for which the participants were not specifically questioned in the participant diary.
Time Frame: 28 days After Vaccination 2 (Day 85 for Groups 1-6; Day 113 for Groups 9 and 10)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 3: Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 4: Ad26.COV2.S 1*10^11 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 5: Ad26.COV2.S 5*10^10 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 9: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 10: Placebo, Placebo, Placebo | Group 1 and 7 Combined | Group 6 and 8 Combined
Number analyzed (Participants) | 81 | 75 | 74 | 81 | 53 | 25 | 141 | 52
Participants | 17 | 15 | 16 | 22 | 10 | 4 | 34 | 9

19. Primary Outcome: Adults of Groups 2 to 5, Group 9-10, 1 and 7 Combined, 6 and 8 Combined: Number of Participants With Serious Adverse Events (SAEs)
Description: SAE is any untoward medical occurrence that at any dose may result in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product.
Time Frame: Up to 1.5 years
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 3: Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 4: Ad26.COV2.S 1*10^11 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 5: Ad26.COV2.S 5*10^10 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 9: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 10: Placebo, Placebo, Placebo | Group 1 and 7 Combined | Group 6 and 8 Combined
Number analyzed (Participants) | 81 | 75 | 74 | 81 | 53 | 25 | 141 | 52
Participants | 1 | 1 | 1 | 2 | 1 | 0 | 7 | 0

20. Primary Outcome: Adults of Groups 2 to 5, Group 9-10, 1 and 7 Combined, 6 and 8 Combined: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: AESIs were significant AEs that were judged to be of special interest because of clinical importance, known or suspected class effects, or based on nonclinical signals. Thrombosis with Thrombocytopenia Syndrome (TTS), a syndrome characterized by a combination of both a thrombotic event and thrombocytopenia, was considered to be an AESI in this study. A suspected TTS case was defined as: Thrombotic events: suspected deep vessel venous or arterial thrombotic events; Thrombocytopenia, defined as platelet count below 150,000/micro liter.
Time Frame: Up to 1.5 years
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 3: Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 4: Ad26.COV2.S 1*10^11 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 5: Ad26.COV2.S 5*10^10 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 9: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 10: Placebo, Placebo, Placebo | Group 1 and 7 Combined | Group 6 and 8 Combined
Number analyzed (Participants) | 37 | 26 | 37 | 44 | 19 | 9 | 141 | 52
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

21. Primary Outcome: Adolescents: Number of Participants With Solicited Local AEs at 7 Days After Vaccination 1
Description: Number of participants with solicited local AEs at 7 days after vaccination 1 were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local AEs were pre-defined local (at the injection site) AEs for which participants were specifically questioned and which were noted by participants in their e-diary for 7 days post vaccination 1 (day of vaccination and the subsequent 7 days). Solicited local AEs included: injection site pain/tenderness, erythema and swelling at the vaccination site.
Time Frame: 7 Days After Vaccination 1 (Day 8)
Population: FAS included all participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A and B Combined: Ad26.COV2.S 2.5*10^10 | Group C: Placebo
Number analyzed (Participants) | 30 | 3
Participants | 29 | 1

22. Primary Outcome: Adolescents: Number of Participants With Solicited Systemic AEs at 7 Days After Vaccination 1
Description: Number of participants with solicited systemic AEs at 7 days after vaccination 1 were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Participants were instructed on how to note signs and symptoms in their diary on a daily basis for 7 days post-vaccination 1 (Day of vaccination1 and the subsequent 7 days) for solicited systemic AEs. Solicited systemic AEs included fatigue, headache, myalgia, nausea and fever (body temperature greater than or equal to [>=] 38 degree Celsius).
Time Frame: 7 Days After Vaccination 1 (Day 8)
Population: FAS included all participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A and B Combined: Ad26.COV2.S 2.5*10^10 | Group C: Placebo
Number analyzed (Participants) | 30 | 3
Participants | 28 | 3

23. Primary Outcome: Adolescents: Number of Participants With Unsolicited AEs at 28 Days After Vaccination 1
Description: Unsolicited AEs were all AEs for which the participants were not specifically questioned in the participant diary.
Time Frame: 28 Days After Vaccination 1 (Day 29)
Population: FAS included all participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A and B Combined: Ad26.COV2.S 2.5*10^10 | Group C: Placebo
Number analyzed (Participants) | 30 | 3
Participants | 12 | 2

24. Primary Outcome: Adolescents: Number of Participants With SAEs (Inclusive Multisystem Inflammatory Syndrome in Children [MIS-C])
Description: SAE was any untoward medical occurrence that at any dose may result in death, was life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a suspected transmission of any infectious agent via a medicinal product.
Time Frame: Up to unblinding date / receipt of a new Covid vaccine (Up to 1.5 years)
Population: FAS included all participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A and B Combined: Ad26.COV2.S 2.5*10^10 | Group C: Placebo
Number analyzed (Participants) | 30 | 3
Participants | 0 | 0

25. Primary Outcome: Adolescents: Number of Participants With AESIs
Description: as for outcome 20
Time Frame: Up to unblinding date / receipt of a new Covid vaccine (Up to 1.5 years)
Population: FAS included all participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A and B Combined: Ad26.COV2.S 2.5*10^10 | Group C: Placebo
Number analyzed (Participants) | 30 | 3
Participants | 0 | 0

26. Secondary Outcome: Adults of Groups 1 to 5, Groups 7 and 9: Percentage of Participants With Serological Response to Vaccination as Measured by VNA Titers 7 Days After Antigen Presentation
Description: Percentage of participants with serological response to vaccination as measured by VNA titers were reported. A participant was considered a responder if at least one of the following conditions was met: 1) The baseline sample value was <=LLOQ and the post-baseline sample was >LLOQ. 2) The baseline sample value was >LLOQ and the post-baseline sample value represented an at least 4-fold (>= 4-fold) increase from the baseline sample value. The lower limit and upper limit of quantification were IC50 of 58 and 12,800 IU/mL, respectively.
Time Frame: 7 days after antigen presentation (Day 176 for Groups 1-5; Day 148 for Group 7; Day 204 for Group 9)
Population: PPI set included all randomized and vaccinated participants with immunogenicity data available excluding participants with major protocol deviations expected to impact immunogenicity outcomes. Due to change in planned analysis, data was not collected and analyzed for Group 7 in this outcome measure. Here "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 2: Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 3: Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 4: Ad26.COV2.S 1*10^11 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 5: Ad26.COV2.S 5*10^10 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 7: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 9: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp
Number analyzed (Participants) | 25 | 33 | 31 | 33 | 27 | 0 | 32
Percentage of participants | 92.0 (74.0) [74.0 to 99.0] | 97.0 (84.2) [84.2 to 99.9] | 83.9 (66.3) [66.3 to 94.5] | 84.8 (68.1) [68.1 to 94.9] | 96.3 (81.0) [81.0 to 99.9] |  | 100.0 (89.1) [89.1 to 100.0]

27. Secondary Outcome: Adults of Groups 1 to 5, Groups 7 and 9: GMTs as Measured by VNA 7 Days After Antigen Presentation
Description: Antibody GMTs as measured by VNA at 7 days after antigen presentation were reported.
Time Frame: 7 days after antigen presentation (Day 176 for Groups 1-5; Day 148 for Group 7; Day 204 for Group 9)
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 2: Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 3: Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 4: Ad26.COV2.S 1*10^11 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 5: Ad26.COV2.S 5*10^10 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 7: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 9: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp
Number analyzed (Participants) | 26 | 33 | 32 | 33 | 28 | 0 | 32
Titer | 318 (207) [207 to 489] | 393 (272) [272 to 568] | 279 (171) [171 to 457] | 275 (182) [182 to 415] | 525 (339) [339 to 814] |  | 616 (462) [462 to 822]

28. Secondary Outcome: Adults of Groups 1 to 5 and Group 9: Percentage of Participants With Serological Response to Vaccination as Measured by S-ELISA 7 Days After Antigen Presentation
Description: as for outcome 2
Time Frame: 7 Days After Antigen Presentation (Day 176 for Groups 1-5 ; Day 204 for Group 9)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 2: Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 3: Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 4: Ad26.COV2.S 1*10^11 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 5: Ad26.COV2.S 5*10^10 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 9: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp
Number analyzed (Participants) | 62 | 62 | 57 | 57 | 57 | 43
Percentage of participants | 100.0 (94.2) [94.2 to 100.0] | 100.0 (94.2) [94.2 to 100.0] | 96.5 (87.9) [87.9 to 99.6] | 100.0 (93.7) [93.7 to 100.0] | 91.2 (80.7) [80.7 to 97.1] | 100.0 (91.8) [91.8 to 100.0]

29. Secondary Outcome: Adults of Group 7: Percentage of Participants With Serological Response to Vaccination as Measured by S-ELISA 7 Days After Antigen Presentation
Description: Percentage of participants with serological response to vaccination as measured by S-ELISA were reported. A participant was considered a responder if at least one of the following conditions was met: 1) The baseline sample value was <=LLOQ and the post-baseline sample was >LLOQ. 2) The baseline sample value was >LLOQ and the post-baseline sample value represented an at least 4-fold (>= 4-fold) increase from the baseline sample value. The lower limit and upper limit of quantification were IC50 of 58 and 12,800 IU/mL. respectively.
Time Frame: Day 148
Population: Modified PPI set included participants who received vaccination 2 within the window (54-64 days).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 7: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp
Number analyzed (Participants) | 31
Percentage of participants | 96.8 [83.3 to 99.9]

30. Secondary Outcome: Adults of Groups 1 to 5 and Group 9: Antibody GMCs as Measured by S-ELISA 7 Days After Antigen Presentation
Description: Antibody GMCs as measured by S-ELISA 7 days after antigen presentation were reported.
Time Frame: 7 Days after Antigen Presentation (Day 176 for Groups 1-5; Day 204 for Group 9)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group 1: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 2: Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 3: Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 4: Ad26.COV2.S 1*10^11 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 5: Ad26.COV2.S 5*10^10 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 9: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp
Number analyzed (Participants) | 65 | 63 | 57 | 58 | 58 | 43
EU/mL | 1146 (904) [904 to 1452] | 1179 (933) [933 to 1490] | 1038 (730) [730 to 1475] | 1024 (721) [721 to 1454] | 1262 (937) [937 to 1702] | 1963 (1514) [1514 to 2545]

31. Secondary Outcome: Adults of Group 7: Antibody GMCs as Measured by S-ELISA 7 Days After Antigen Presentation
Description: Antibody GMCs as measured by S-ELISA 7 days after antigen presentation were reported.
Time Frame: Day 148
Population: Modified PPI set included participants who received vaccination 2 within the window (54-64 days).
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group 7: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp
Number analyzed (Participants) | 31
EU/mL | 1141 [721 to 1805]

32. Secondary Outcome: Adults of Groups 2 to 5, Group 9-10, 1 and 7 Combined, 6 and 8 Combined: Number of Participants With Solicited Local AEs at 7 Days After Antigen Presentation
Description: Number of participants with solicited local AEs at 7 days after antigen presentation were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local AEs were pre-defined local (at the injection site) AEs for which participants were specifically questioned and which were noted by participants in their e-diary for 7 days after antigen presentation (day of antigen presentation and the subsequent 7 days). Solicited local AEs included: injection site pain/tenderness, erythema and swelling at the vaccination site.
Time Frame: 7 Days After Antigen Presentation (Day 176 for Groups 2-5, Groups 1 and 7 combined, Groups 6 and 8 combined; Day 204 for Group 9 and 10)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 3: Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 4: Ad26.COV2.S 1*10^11 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 5: Ad26.COV2.S 5*10^10 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 9: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 10: Placebo, Placebo, Placebo | Group 1 and 7 Combined | Group 6 and 8 Combined
Number analyzed (Participants) | 69 | 68 | 68 | 74 | 47 | 18 | 127 | 44
Participants | 28 | 29 | 31 | 35 | 16 | 2 | 50 | 1

33. Secondary Outcome: Adults of Groups 2 to 5, Group 9-10, 1 and 7 Combined, 6 and 8 Combined: Number of Participants With Solicited Systemic AEs at 7 Days After Antigen Presentation
Description: Number of participants with solicited systemic AEs at 7 days after antigen presentation were reported. An AE was any untoward medical occurrence in a Participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Participants were instructed on how to note signs and symptoms in their diary on a daily basis for 7 days after antigen presentation (Day of antigen presentation and the subsequent 7 days) for solicited systemic AEs. Solicited systemic AEs included fatigue, headache, myalgia, nausea and fever (body temperature greater than or equal to [>=] 38 degree Celsius).
Time Frame: as for outcome 32
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 3: Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 4: Ad26.COV2.S 1*10^11 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 5: Ad26.COV2.S 5*10^10 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 9: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 10: Placebo, Placebo, Placebo | Group 1 and 7 Combined | Group 6 and 8 Combined
Number analyzed (Participants) | 69 | 68 | 68 | 74 | 47 | 18 | 127 | 44
Participants | 30 | 24 | 23 | 28 | 15 | 4 | 51 | 10

34. Secondary Outcome: Adults of Groups 2 to 5, Group 9-10, 1 and 7 Combined, 6 and 8 Combined: Number of Participants With Unsolicited AEs at 28 Days After Antigen Presentation
Description: Unsolicited AEs were all AEs for which the participants were not specifically questioned in the participants diary.
Time Frame: 28 Days After Antigen Presentation (Day 197 for Groups 2-5, Groups 1 and 7 combined, Groups 6 and 8 combined; Day 225 for Group 9 and 10)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 3: Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 4: Ad26.COV2.S 1*10^11 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 5: Ad26.COV2.S 5*10^10 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 9: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 10: Placebo, Placebo, Placebo | Group 1 and 7 Combined | Group 6 and 8 Combined
Number analyzed (Participants) | 69 | 68 | 68 | 74 | 47 | 18 | 127 | 44
Participants | 10 | 7 | 6 | 12 | 6 | 4 | 15 | 4

35. Secondary Outcome: Adults of Groups 2 to 5, Group 9-10, 1 and 7 Combined, 6 and 8 Combined: Number of Participants With SAEs After Antigen Presentation
Description: as for outcome 19
Time Frame: After antigen presentation until end of study (Day 170 up to 1.5 years for Groups 2-5, Groups 1 and 7 combined, Groups 6 and 8 combined; Day 198 up to 1.5 years for Group 9 and 10)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 3: Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 4: Ad26.COV2.S 1*10^11 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 5: Ad26.COV2.S 5*10^10 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 9: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 10: Placebo, Placebo, Placebo | Group 1 and 7 Combined | Group 6 and 8 Combined
Number analyzed (Participants) | 69 | 68 | 68 | 74 | 47 | 18 | 127 | 44
Participants | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0

36. Secondary Outcome: Adults of Groups 2 to 5, Group 9-10, 1 and 7 Combined, 6 and 8 Combined: Number of Participants With AESIs After Antigen Presentation
Description: AESIs were significant AEs that were judged to be of special interest because of clinical importance, known or suspected class effects, or based on nonclinical signals. Thrombosis with Thrombocytopenia Syndrome (TTS), a syndrome characterized by a combination of both a thrombotic event and thrombocytopenia, is considered to be an AESI in this study. A suspected TTS case was defined as: Thrombotic events: suspected deep vessel venous or arterial thrombotic events; Thrombocytopenia, defined as platelet count below 150,000/micro liter.
Time Frame: as for outcome 35
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 3: Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 4: Ad26.COV2.S 1*10^11 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 5: Ad26.COV2.S 5*10^10 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 9: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 10: Placebo, Placebo, Placebo | Group 1 and 7 Combined | Group 6 and 8 Combined
Number analyzed (Participants) | 69 | 68 | 68 | 74 | 47 | 18 | 127 | 44
Participants | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

37. Secondary Outcome: Adults Groups 1 to 6: Percentage of Participants With Neutralizing Antibody Titers to the Wild-type SARS-CoV-2 Virus Expressing S-protein as Measured by VNA
Description: Percentage of participants with neutralizing antibody titers to the wild-type SARS-CoV-2 virus expressing S-protein as measured by VNA were reported.
Time Frame: Days 197 and 393
Population: PPI set was analyzed. Here, 'N' (Overall number of participants analyzed) signifies participants evaluated for this outcome measure. Here 'n' (number analyzed) signifies number of participants evaluable at specified time points.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 2: Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 3: Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 4: Ad26.COV2.S 1*10^11 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 5: Ad26.COV2.S 5*10^10 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 6: Placebo, Placebo, Placebo
Number analyzed (Participants) | 29 | 31 | 29 | 31 | 26 | 12
Percentage of participants
  Day 197: number analyzed (Participants) | 26 | 31 | 29 | 31 | 26 | 12
  Day 197 | 100.0 [86.8 to 100.0] | 100.0 [88.8 to 100.0] | 96.6 [82.2 to 99.9] | 96.8 [83.3 to 99.9] | 80.8 [60.6 to 93.4] | 0.0 [0.0 to 26.5]
  Day 393: number analyzed (Participants) | 29 | 21 | 19 | 30 | 26 | 0
  Day 393 | 93.1 [77.2 to 99.2] | 95.2 [76.2 to 99.9] | 84.2 [60.4 to 96.6] | 80.0 [61.4 to 92.3] | 92.0 [74.0 to 99.0] |

38. Secondary Outcome: Adults Group 9 and 10: Percentage of Participants With Neutralizing Antibody Titers to the Wild-type SARS-CoV-2 Virus Expressing S-protein as Measured by VNA
Description: as for outcome 37
Time Frame: Days 225 and 421
Population: as for outcome 37
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 9: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 10: Placebo, Placebo, Placebo
Number analyzed (Participants) | 31 | 10
Percentage of participants
  Day 225: number analyzed (Participants) | 29 | 10
  Day 225 | 100.0 [88.1 to 100.0] | 0.0 [0.0 to 30.8]
  Day 421: number analyzed (Participants) | 31 | 1
  Day 421 | 100.0 [88.8 to 100.0] | 0.0 [0.0 to 97.5]

39. Secondary Outcome: Adults Groups 1 to 6: Percentage of Participants With Binding Antibody Titers to SARS-CoV-2 or Individual SARS-CoV-2 Proteins
Description: Percentage of participants with binding antibody titers to SARS-CoV-2 or individual SARS-CoV-2 proteins were reported.
Time Frame: Days 197 and 393
Population: as for outcome 37
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 2: Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 3: Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 4: Ad26.COV2.S 1*10^11 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 5: Ad26.COV2.S 5*10^10 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 6: Placebo, Placebo, Placebo
Number analyzed (Participants) | 63 | 60 | 55 | 55 | 56 | 16
Percentage of participants
  Day 197: number analyzed (Participants) | 62 | 60 | 55 | 55 | 56 | 16
  Day 197 | 100.0 [94.2 to 100.0] | 100.0 [94.0 to 100.0] | 98.2 [90.3 to 100.0] | 100.0 [93.5 to 100.0] | 98.2 [90.4 to 100.0] | 0.0 [0.0 to 20.6]
  Day 393: number analyzed (Participants) | 63 | 33 | 28 | 51 | 51 | 0
  Day 393 | 100.0 [94.3 to 100.0] | 100.0 [89.4 to 100.0] | 85.7 [67.3 to 96.0] | 92.2 [81.1 to 97.8] | 98.0 [89.6 to 100.0] |

40. Secondary Outcome: Adults of Groups 9 and 10: Percentage of Participants With Binding Antibody Titers to SARS-CoV-2 or Individual SARS-CoV-2 Proteins
Description: Percentage of participants with binding antibody titers to SARS-CoV-2 or individual SARS-CoV-2 proteins were reported.
Time Frame: Days 225 and 421
Population: as for outcome 37
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 9: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 10: Placebo, Placebo, Placebo
Number analyzed (Participants) | 39 | 14
Percentage of participants
  Day 225: number analyzed (Participants) | 37 | 14
  Day 225 | 100.0 [90.5 to 100.0] | 0.0 [0.0 to 23.2]
  Day 421: number analyzed (Participants) | 39 | 1
  Day 421 | 97.4 [86.5 to 99.9] | 0.0 [0.0 to 97.5]

41. Secondary Outcome: Adolescents: Percentage of Participants With Serological Response to Vaccination as Measured by VNA Titers 28 Days After Vaccination 1 (Day 29)
Description: as for outcome 5
Time Frame: 28 Days After Vaccination 1 (Day 29)
Population: PPI set included all randomized and vaccinated participants with immunogenicity data available excluding participants with major protocol deviations expected to impact immunogenicity outcomes. Samples obtained after missed vaccinations or participants with natural SARS-CoV-2 infection (defined as a positive PCR test or positive N-serology) occurring after screening were excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group A and B Combined: Ad26.COV2.S 2.5*10^10 | Group C: Placebo
Number analyzed (Participants) | 27 | 3
Percentage of participants | 100.0 (87.2) [87.2 to 100.0] | 0.0 (0.0) [0.0 to 70.8]

42. Secondary Outcome: Adolescents: Percentage of Participants With Serological Response to Vaccination as Measured by S-ELISA 28 Days After Vaccination 1 (Day 29)
Description: as for outcome 2
Time Frame: 28 Days After Vaccination 1 (Day 29)
Population: as for outcome 41
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group A and B Combined: Ad26.COV2.S 2.5*10^10 | Group C: Placebo
Number analyzed (Participants) | 27 | 3
Percentage of participants | 100.0 (86.8) [86.8 to 100.0] | 0.0 (0.0) [0.0 to 70.8]

43. Secondary Outcome: Adolescents: Antibody GMTs as Measured by VNA at 28 Days After Vaccination 1
Description: Antibody GMTs as measured by VNA at 28 days after vaccination 1 (Day 29) were reported. LLOQ was 58 IU/mL
Time Frame: 28 days After Vaccination 1 (Day 29)
Population: as for outcome 41
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group A and B Combined: Ad26.COV2.S 2.5*10^10 | Group C: Placebo
Number analyzed (Participants) | 27 | 3
Titer | 305 [245 to 378] | NA [NA to NA] — 'Geometric mean' and 95% confidence interval could not be estimated as the analyzed values were below the LLOQ.

44. Secondary Outcome: Adolescents: Antibody GMCs as Measured by S-ELISA 28 Days After Vaccination 1
Description: Antibody GMCs as measured by S-ELISA 28 days after vaccination was reported. LLOQ was 58 IU/mL
Time Frame: 28 days After Vaccination 1 (Day 29)
Population: as for outcome 41
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Group A and B Combined: Ad26.COV2.S 2.5*10^10 | Group C: Placebo
Number analyzed (Participants) | 27 | 3
EU/mL | 682 [506 to 920] | NA [NA to NA] — "Geometric Mean" and "95% Confidence Interval" data could not be estimated as the analyzed value were below the LLOQ.

45. Secondary Outcome: Adolescents: Neutralizing Antibody Titers to the Wild-type SARS-CoV-2 Virus Expressing S Protein as Measured by VNA
Description: Neutralizing antibody titers to the Wild-type SARS-CoV-2 virus expressing S protein measured by VNA was reported. LLOQ was 58 IU/mL.
Time Frame: Days 57, 85 and 169
Population: PPI set included all randomized and vaccinated participants with immunogenicity data available excluding participants with major protocol deviations expected to impact immunogenicity outcomes. Samples obtained after missed vaccinations or participants with natural SARS-CoV-2 infection (defined as a positive PCR test or positive N-serology) occurring after screening were excluded from the analysis. "Number analyzed" signifies participants evaluable at specified time points.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group A and B Combined: Ad26.COV2.S 2.5*10^10 | Group C: Placebo
Number analyzed (Participants) | 27 | 3
Titer
  Day 57 | 323 [262 to 399] | NA [NA to NA] — "Geometric Mean" and "95% Confidence Interval" data could not be estimated as the analyzed value were below the LLOQ.
  Day 85: number analyzed (Participants) | 22 | 3
  Day 85 | 306 [227 to 413] | NA [NA to NA] — "Geometric Mean" and "95% Confidence Interval" data could not be estimated as the analyzed value were below the LLOQ.
  Day 169: number analyzed (Participants) | 15 | 0
  Day 169 | 342 [219 to 532] |

46. Secondary Outcome: Adolescents: Binding Antibody Titers to SARS-CoV-2 or Individual SARS-CoV-2 Proteins as Measured by ELISA
Description: Binding antibody titers to SARS-CoV-2 or individual SARS-CoV-2 proteins as measured by ELISA was reported. LLOQ was 58 IU/mL.
Time Frame: Days 57, 85, 169
Population: as for outcome 45
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group A and B Combined: Ad26.COV2.S 2.5*10^10 | Group C: Placebo
Number analyzed (Participants) | 27 | 3
Titer
  Day 57 | 770 [593 to 1000] | NA [NA to NA] — "Geometric Mean" and "95% Confidence Interval" data could not be estimated as the analyzed value were below the LLOQ.
  Day 85: number analyzed (Participants) | 22 | 3
  Day 85 | 773 [547 to 1093] | NA [NA to NA] — "Geometric Mean" and "95% Confidence Interval" data could not be estimated as the analyzed value were below the LLOQ.
  Day 169: number analyzed (Participants) | 15 | 0
  Day 169 | 796 [449 to 1411] |

47. Secondary Outcome: Adults: Percentage of Participants With Serological Response to Vaccination as Measured by S-ELISA 7 Days After Antigen Presentation
Description: as for outcome 2
Time Frame: 7 Days After Antigen Presentation (Day 176 for Groups 1-5 ; Day 204 for Group 9)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 2: Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 3: Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 4: Ad26.COV2.S 1*10^11 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 5: Ad26.COV2.S 5*10^10 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 9: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp
Number analyzed (Participants) | 62 | 62 | 57 | 57 | 57 | 43
Percentage of participants | 100.0 (94.2) [94.2 to 100.0] | 100.0 (94.2) [94.2 to 100.0] | 96.5 (87.9) [87.9 to 99.6] | 100.0 (93.7) [93.7 to 100.0] | 91.2 (80.7) [80.7 to 97.1] | 100.0 (91.8) [91.8 to 100.0]

ADVERSE EVENTS:
Time Frame: Up to 1.5 years
Description: FAS included all participants with at least one vaccine administration documented. 55 participants from group 7 and 26 participants from group 8 with vaccination 2 delayed due to study pause were analyzed with groups 1 and 6 respectively. However, 1 participant in group 7 and 1 participant in group 8 received the second vaccination as scheduled (28 days after first vaccination). Therefore, adverse events for these 2 participants were included in Groups 7 and 8 reporting arms.
Arm/Group | Group 1: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 2: Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 3: Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 4: Ad26.COV2.S 1*10^11 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 5: Ad26.COV2.S 5*10^10 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp | Group 6: Placebo, Placebo, Placebo | Group 7: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 8: Placebo, Placebo, Placebo | Group 9: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp | Group 10: Placebo, Placebo, Placebo | Group A and B Combined: Ad26.COV2.S 2.5*10^10 | Group C: Placebo
All-Cause Mortality (participants affected / at risk) | 0/141 | 1/81 | 0/75 | 0/74 | 0/81 | 0/52 | 0/1 | 0/1 | 0/53 | 0/25 | 0/30 | 0/3
Serious Adverse Events (participants affected / at risk) | 7/141 | 1/81 | 1/75 | 1/74 | 2/81 | 0/52 | 0/1 | 0/1 | 1/53 | 0/25 | 0/30 | 0/3
Other Adverse Events (participants affected / at risk) | 35/141 | 24/81 | 20/75 | 20/74 | 33/81 | 11/52 | 0/1 | 0/1 | 16/53 | 9/25 | 11/30 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp (N=141) | Group 2: Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp (N=81) | Group 3: Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp (N=75) | Group 4: Ad26.COV2.S 1*10^11 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp (N=74) | Group 5: Ad26.COV2.S 5*10^10 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp (N=81) | Group 6: Placebo, Placebo, Placebo (N=52) | Group 7: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp (N=1) | Group 8: Placebo, Placebo, Placebo (N=1) | Group 9: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp (N=53) | Group 10: Placebo, Placebo, Placebo (N=25) | Group A and B Combined: Ad26.COV2.S 2.5*10^10 (N=30) | Group C: Placebo (N=3)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic Cyst (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic Candida (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrospinal Fluid Leakage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp (N=141) | Group 2: Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 2.5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp (N=81) | Group 3: Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp, Ad26.COV2.S 1.25*10^10 vp (N=75) | Group 4: Ad26.COV2.S 1*10^11 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp (N=74) | Group 5: Ad26.COV2.S 5*10^10 vp, Placebo, Ad26.COV2.S 1.25*10^10 vp (N=81) | Group 6: Placebo, Placebo, Placebo (N=52) | Group 7: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp (N=1) | Group 8: Placebo, Placebo, Placebo (N=1) | Group 9: Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 5*10^10 vp, Ad26.COV2.S 1.25*10^10 vp (N=53) | Group 10: Placebo, Placebo, Placebo (N=25) | Group A and B Combined: Ad26.COV2.S 2.5*10^10 (N=30) | Group C: Placebo (N=3)
Eye Pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (3)
Chills (General disorders) | 5 (6) | 5 (6) | 1 (1) | 2 (2) | 4 (4) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Fatigue (General disorders) | 5 (6) | 5 (7) | 2 (2) | 4 (5) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (2)
Covid-19 (Infections and infestations) | 3 (5) | 3 (3) | 4 (5) | 0 (0) | 4 (4) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 7 (8) | 0 (0)
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (5) | 1 (1) | 7 (7) | 5 (6) | 8 (8) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2) | 2 (2) | 4 (5) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 18 (18) | 11 (17) | 8 (10) | 11 (14) | 15 (19) | 7 (9) | 0 (0) | 0 (0) | 9 (12) | 6 (9) | 0 (0) | 0 (0)
Premenstrual Pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4) | 2 (3) | 3 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 1 (1) | 4 (5) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 3 (3) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 5 (6) | 4 (5) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (3):
  • Study Protocol (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/53/NCT04535453/Prot_001.pdf
  • Statistical Analysis Plan (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/53/NCT04535453/SAP_002.pdf
  • Informed Consent Form (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/53/NCT04535453/ICF_003.pdf